CLINICAL TRIAL: NCT00326794
Title: Effectiveness at 3 Months of Immediate Shoulder Mobilisation Versus Conventional Immobilisation for Impacted Nonsurgically Treated Proximal Humerus Fracture: a Randomised Controlled Trial.
Brief Title: Efficacy of Shoulder Mobilisation Versus Conventional Immobilisation for Nonsurgically Proximal Humerus Fracture
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P011022
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2006-05-17 (Estimated); Status verified 2005-06

CONDITIONS: Shoulder Fracture
Keywords: Nonsurgical proximal humerus fracture; Rehabilitation; Physiotherapy; randomised controlled trial
MeSH Terms: conditions — Shoulder Fractures | interventions — Rehabilitation

INTERVENTIONS:
Procedure: mobilisation (rehabilitation)

SUMMARY:
Background: Nonsurgical proximal humerus fracture is common, causing prolonged disability, for which the time to begin rehabilitation is not well determined. We assessed the feasibility and efficacy of early (within 3 days'after fracture) mobilisation of the shoulder compared with conventional 3-week immobilization followed by physiotherapy.

DETAILED DESCRIPTION:
Methods: We randomly assigned 74 patients with impacted nonsurgically treated proximal humerus fracture to receive early passive mobilisation or conventional-treatment. The primary outcome was functional assessment of the shoulder (Constant score) at 3 months. Secondary outcomes were functional assessment at 6 weeks and at 6 months, change in pain (on a visual analogue scale) and passive range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Impacted nonsurgically treated proximal humerus fracture
* Patients over the age 20

Exclusion Criteria:

* Pre-existing shoulder pathology
* Neurological disorders of the upper limbs
* Indication for surgery of the shoulder
* Combined polytrauma
* Difficulties with language or comprehension to understand a rehabilitation program and information

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76
Dates: Start 2002-10; Study Completion 2005-09

PRIMARY OUTCOMES:
The primary outcome was functional assessment of the shoulder (Constant score) at 3 months.

SECONDARY OUTCOMES:
Functional assessment at 6 weeks and at 6 months
Change in pain (on a visual analogue scale)at 6 weeks, 3 months and at 6 months
Passive range of motion at 6 weeks, 3 months and at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Martine Lefevre-colau, MDPhD, Principal Investigator — APHP
Locations (1):
- Hopital Cochin, Paris, France